CLINICAL TRIAL: NCT06492434
Title: Enhancing Community Participation Outcomes Among Young Adults With Serious Mental Illnesses Through Peer-Delivered Decision Support
Brief Title: Enhancing Community Participation Through Peer-Delivered Decision Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 270034; 90IFRE0068 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Severe Mental Disorder
Keywords: Peer specialists, Decision Support Techniques, Young Adult
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer decision coaching arm (Experimental): All participants will engage in the Peer Decision Coaching intervention.
  Interventions: Behavioral: Peer decision coaching

INTERVENTIONS:
Behavioral: Peer decision coaching — Peer Decision Coaching is a brief, personalized intervention grounded in evidence-based decision- and peer support principles. During the intervention, a trained peer specialist supports the young person in identifying a decision related to community participation that they need to make, such as whether to work or go to school, helping them address decision-making needs, and assisting them with developing and implementing a decision-making plan. Ultimately, the intervention aims to support young people in pursuing their community participation interests and goals.

SUMMARY:
The purpose of this study is to pilot test a peer-delivered decision support intervention ("peer decision coaching") designed to enhance decision-making about community participation among young adults with serious mental illness (SMI).

DETAILED DESCRIPTION:
The overarching goal of this study is to pilot test a peer-delivered decision support intervention ("peer decision coaching") designed to enhance decision-making about community participation among young adults with serious mental illnesses (SMI). We will use a single-group, pre-post, convergent mixed methods design to explore implementation and whether and how the intervention impacts decision-making and community participation outcomes. We will aim to recruit 40 participants in this intervention study. This design will enable us to link themes regarding participants' experience of the intervention with quantitative measures of decision-making and community participation.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age;
* Experiencing a SMI, as determined by: (a) self-reported psychiatric diagnosis of schizophrenia-spectrum or major affective disorder, and (b) self-reported current or past functional impairment due to experiencing mental health challenges in one or more major life areas (i.e., work school, social activities)
* Able to identify at least 2 areas of community participation that individuals want to be doing more in in the next 6 months
* Current sufficiency of community participation (i.e., number of important participation areas done enough / number of important participation areas) of 50% or less.

Exclusion Criteria:

* Unable to provide informed consent, as assessed by research staff using an active recall method
* limited ability to act on decisions due to self-reported legal, residential, or guardianship restrictions.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Change in decisional conflict scale | Baseline, through intervention completion (up to 3 months)
  The Factors Contributing to Uncertainty subscale of the Decisional Conflict Scale measures decision-making needs. Possible scores range from 0 to 36, with higher scores indicating a worse outcome.
Change in decision self-efficacy scale | Baseline, through intervention completion (up to 3 months)
  The Decision Self-Efficacy Scale assesses confidence in making an informed choice. Possible scores range from 0 to 44, with higher scores indicating a better outcome.
Decision-making behaviors at post-intervention | Post-intervention (up to 3 months post-baseline)
  Number of behaviors (range: 0-6) endorsed on Decision-Making Behaviors scale at post-intervention.
Decision Satisfaction Scale Score at post-intervention | Post-intervention (up to 3 months post-baseline)
  The Decision Satisfaction Scale assesses a person's satisfaction with a health decision. Possible scores range from 6-30, with higher scores indicating a better outcome.
Change in Temple University Community Participation Measure (sufficiency) | Baseline, through intervention completion (up to 3 months)
  Sufficiency scores on the Temple University Community Participation Measure assess how satisfied individuals are with their amount of community participation in areas that are important to them. Possible scores range from 0-100, with higher scores indicating a better outcome.
Change in Temple University Community Participation Measure (breadth ratio) | Baseline, through intervention completion (up to 3 months)
  Breadth ratio scores on the Temple University Participation Measure assess breadth of participation in areas considered important to a person. Possible scores range from 0-100, with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Thomas, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Temple University, Philadelphia, Pennsylvania
  - Copeland Center for Wellness and Recovery, Brattleboro, Vermont